CLINICAL TRIAL: NCT06909084
Title: Comparison of Outcome of Myringotomy With or Without Ventilation Tube in Children With Glue Ears
Brief Title: Hearing Improvement After Making a Hole Surgically in Eardrum With or Without Ventilation Tube in Children With Glue Ears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allama Iqbal Teaching Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Mudasir Abbas, Principal Investigator, Allama Iqbal Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1317-1361
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Otitis Media With Effusion in Children; Hearing Loss
Keywords: Otitis Media with Effusion; Hearing Loss; Children; Middle ear Ventilation
MeSH Terms: conditions — Hearing Loss; Otitis Media with Effusion | interventions — Middle Ear Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Myringotomy with Ventilation tube (Experimental): A tympanostomy tube (Shepard tube) of appropriate size will be placed in the incision and canal will be packed with bismuth iodoform paraffin paste (BIPP)
  Interventions: Procedure: Myringotomy with ventilation tube
- Myringotomy alone (Active Comparator): Incision in the eardrum (myringotomy) will be made. Middle ear canal will be cleaned after draining the fluid and the canal will be packed with bismuth iodoform paraffin paste (BIPP)
  Interventions: Procedure: Myringotomy alone

INTERVENTIONS:
Procedure: Myringotomy with ventilation tube — Under microscope tympanic membrane was visualized after cleaning the external auditory canal and myringotomy incision was given with the help of myringotome in anteroinferior quadrant of tympanic membrane. Secretions from middle ear were drained by suction. A tympanostomy tube (Shepard tube) of appropriate size was placed in the incision and canal was packed with bismuth iodoform paraffin paste which was removed after 24 hours.
  Arms: Myringotomy with Ventilation tube
Procedure: Myringotomy alone — Under microscope tympanic membrane was visualized after cleaning the external auditory canal and myringotomy incision was given with the help of myringotome in anteroinferior quadrant of tympanic membrane. Secretions from middle ear were drained by suction. NO FURTHER PROCEDURE WAS DONE and canal was packed with bismuth iodoform paraffin paste which was removed after 24 hours.
  Arms: Myringotomy alone

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of myringotomy with ventilation tube insertion to myringotomy alone in improving hearing in children with glue ear.

The main question it aims to answer is:

Does adding a ventilation tube to myringotomy lead to greater improvement in hearing compared to myringotomy alone? Researchers will compare these two surgical techniques to determine which offers better outcomes for children with otitis media with effusion.

The Participants will:

1. Have their hearing evaluated before surgery
2. Undergo either myringotomy with ventilation tube insertion or myringotomy alone
3. Have their hearing evaluated at follow-up visits at 2 weeks, 1 month, and 3 months post-operatively

ELIGIBILITY:
Inclusion Criteria:

* cases of otitis media with effusion
* more than 20 decibel (dB) conductive hearing loss on pure tone audiometry
* non-responder to medical treatment after three months of medical treatment

Exclusion Criteria:

* Children having recurrent otitis media
* Discharging ears
* History of bleeding disorder

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Improvement in hearing | Before and Three months post operatively
  The degree of hearing loss (dB) on pure tone audiometry was done before and after surgical procedure. Improvement in hearing level was labelled if there was decrease in hearing loss of 25% from baseline.

SECONDARY OUTCOMES:
Hearing Loss (dB) | Before and Three months post operatively
  All patients underwent pure tone audiometry for assessment of hearing loss (dB)
Degree of Hearing Loss | Before and Three months post operatively
  The degree of hearing loss (dB) on pure tone audiometry was done before and after surgical procedure. Degree of hearing loss was labelled as mild (20-40 dB), moderate (40-60 dB) and severe (60-80 dB).

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sharbaz Hussain Khosa, FCPS, Study Chair — Allama Iqbal Teaching Hospital Dera Ghazi Khan
Locations (1):
- Allama Iqbal Teaching Hospital Dera Ghazi Khan, Dera Ghazi Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) might not be shared because it contains sensitive personal health information. Sharing such data could compromise participant confidentiality and privacy, and may conflict with ethical guidelines, informed consent, and regulatory requirements.